CLINICAL TRIAL: NCT06168773
Title: Combination of Haloperidol and Magnesium for Delirium Prevention in Critically Ill Elderly Patients After Elective Major Surgery
Brief Title: Combination of Haloperidol and Magnesium for Delirium Prevention in Critically Ill Elderly
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Salah Eldin Mahmoud Badre, Associate Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU R168/2021
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Delirium in Old Age
MeSH Terms: interventions — Haloperidol; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: Group I (number of patients = 45): will receive 1 mg haloperidol intravenously 3 times daily and magnesium sulfate 4 g intravenous infusion (IVI) in 1st day (diluted in 50 ml D5W over 24 hours) then 2g IVI over 24 hours (diluted in 50 ml D5W over 24 hours) for 3 days postoperatively starting the first dose 2- 4 hours after surgery. If the first prophylactic dose is delayed for more than 4 hours post admission, patient is excluded from the study.
  Group II (number of patients= 45): will receive 1 mg haloperidol intravenously 3 times daily and 50 ml of D5W IVI infusion over 24 hours for 4 days postoperatively starting the first dose 2- 4 hours after surgery.
  Group III (number of patients = 45): will receive 1 mL 0.9% of sodium chloride intravenously 3 times daily and 50 ml of D5W IVI infusion for 4 days postoperatively starting the first dose 2- 4 hours after surgery.
Who Masked: Participant, Investigator
Masking Description: prospective randomized double-blind placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group I (number of patients = 45): (Experimental): will receive 1 mg haloperidol intravenously 3 times daily and magnesium sulfate 4 g intravenous infusion (IVI) in 1st day (diluted in 50 ml D5W over 24 hours) then 2g IVI over 24 hours (diluted in 50 ml D5W over 24 hours) for 3 days postoperatively starting the first dose 2- 4 hours after surgery. If the first prophylactic dose is delayed for more than 4 hours post admission, patient is excluded from the study.
  Interventions: Drug: Haloperidol Injection
- Group II (number of patients= 45): (Experimental): will receive 1 mg haloperidol intravenously 3 times daily and 50 ml of D5W IVI infusion over 24 hours for 4 days postoperatively starting the first dose 2- 4 hours after surgery.
  Interventions: Drug: Haloperidol Injection
- Group III (number of patients = 45) (Placebo Comparator): will receive 1 mL 0.9% of sodium chloride intravenously 3 times daily and 50 ml of D5W IVI infusion for 4 days postoperatively starting the first dose 2- 4 hours after surgery.
  Interventions: Drug: Haloperidol Injection

INTERVENTIONS:
Drug: Haloperidol Injection — to evaluate the efficacy and safety of short-term intravenous combination of low-dose haloperidol and magnesium for delirium prevention in critically ill elderly patients after elective major surgery.
  Other Names: Magnesium Sulphate

SUMMARY:
Objective: The aim of this randomized double blinded study is to investigate the effectiveness and safety of the prophylactic use of haloperidol with or without magnesium (Mg) for delirium in high risk elderly patients postoperatively.

Patients and methods: 135 patients aged ≥ 65< 80 years old with PRE-DELIRIC Score 50% or more (20) were admitted to the ICU non-intubated following major non cardiac surgeries randomized into 3 groups, Group I received 1 mg haloperidol intravenously 3 times daily and magnesium sulfate 4 g intravenous infusion (IVI) in 1st day (diluted in 50 ml D5W over 24 hours) then 2g IVI over 24 hours (diluted in 50 ml D5W over 24 hours) for 3 days, Group II received 1 mg haloperidol intravenously 3 times ,Group III received 1 mL 0.9% of sodium chloride intravenously 3 times daily. The primary outcome of the study will be the incidence of delirium.

DETAILED DESCRIPTION:
This prospective randomized double-blind placebo-controlled study will be conducted in Ain Shams university surgical ICU on 135 patients aged ≥ 65< 80 years old with PRE-DELIRIC Score 50% or more (20) who are admitted to the ICU non-intubated following major non cardiac surgeries and anticipated intensive care unit (ICU) stay of at least 2 days as estimated by the attending intensivist after the approval of the research ethical committee and obtaining patients' or patients ' relatives written informed consent.

The study medications are continued until ICU discharge or until delirium occurred. In the latter case, study medications are stopped, and patients could be treated with dexmedetomidine.

For delirium prevention non-pharmacological interventions are also implemented like early mobilization, improving patient circadian rhythm, noise reduction are parts of the daily ICU care.

Patients will receive fentanyl infusion for analgesia. Those patients achieving a RASS score of ± 1 or 0 are monitored daily for delirium using the Confusion Assessment Method for the ICU (CAM-ICU). Patients are diagnosed with delirium if they have at least 1 positive CAM-ICU without RASS -4/-5 during a complete day. Clinicians collecting data on delirium are all experienced in delirium assessment using the CAM-ICU. All patients are screened at least three times daily, and more often if required.

ELIGIBILITY:
Inclusion Criteria:

- PRE-DELIRIC Score 50% or more (20) who are admitted to the ICU non-intubated following major non cardiac surgeries and anticipated intensive care unit (ICU) stay of at least 2 days as estimated by the attending intensivist

Exclusion Criteria:

* sustained RASS of -4/-5 during the complete ICU admission
* primary neurologic event/injury with GCS ≤ 9 during the first 48 hours of ICU
* delirium prior to inclusion, Parkinson disease, dementia, alcohol abuse, an acute neurological condition, history of a psychiatric disease and use of antipsychotic agents
* history of clinically relevant ventricular arrhythmia in the last 12 months, QTc time of at least 500 milliseconds
* recent MI or cardiac decompensation, 2nd or 3rd AV block
* Known allergy or intolerance to haloperidol or magnesium sulphate.
* 80 years or older, had a body weight of 50 kg or less, or had liver failure (serum bilirubin level >2.9 mg/dL) or serum creatinine level >150 μmol/L
* Intubated patients at the time of ICU admission.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 135 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
the incidence of delirium | for 3 days postoperatively starting the first dose 2- 4 hours after surgery.
  Patients will receive fentanyl infusion for analgesia. Those patients achieving a RASS score of ± 1 or 0 are monitored daily for delirium using the Confusion Assessment Method for the ICU (CAM-ICU). Patients are diagnosed with delirium if they have at least 1 positive CAM-ICU without RASS -4/-5 during a complete day.

SECONDARY OUTCOMES:
The occurrence of extra-pyramidal symptoms. | during 3 days postoperative
  The occurrence of extra-pyramidal symptoms, such as dystonia, tremor, myoclonus, tics, rigidity, and akathisia.

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
share the protocol